CLINICAL TRIAL: NCT02541682
Title: Assessment of the Relationship Between Affective Temperament and the Severity of Nausea and Vomiting in Early Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemalpasa Government Hospital (Other)
Responsible Party: Principal Investigator, ALI BAHADIRLI, Specialist, Mustafa Kemalpasa Government Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TUTF-GOKAEK 2013/50
Record Dates: First submitted 2015-08-30; First posted 2015-09-04 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Hyperemesis Gravidarum; Temperament; Morning Sickness
MeSH Terms: conditions — Hyperemesis Gravidarum; Morning Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Other): Participants who have PUQE ( Pregnancy Unique Quantification of Emesis scoring index) score equal to 3 and showing no symptom of nausea and/or vomiting during the three control visits. Control visits are performed a month apart.
  Interventions: Other: TEMPS-A (Temperament Evaluation of Memphis, Pisa, Paris and San Diego Auto-questionnaire)
- Mild nausea and vomiting of pregnancy (Other): Participants who have maximum PUQE ( Pregnancy Unique Quantification of Emesis scoring index) score equal to 4-6 during the three control visits. Control visits are performed a month apart.
  Interventions: Other: TEMPS-A (Temperament Evaluation of Memphis, Pisa, Paris and San Diego Auto-questionnaire)
- Moderate nausea and vomiting of pregnancy (Other): Participants who have maximum PUQE ( Pregnancy Unique Quantification of Emesis scoring index) score equal to 7-12 during the three control visits. Control visits are performed a month apart.
  Interventions: Other: TEMPS-A (Temperament Evaluation of Memphis, Pisa, Paris and San Diego Auto-questionnaire)
- Severe nausea and vomiting of pregnancy (Other): Participants who have maximum PUQE ( Pregnancy Unique Quantification of Emesis scoring index) score equal to 13-15 during the three control visits. Control visits are performed a month apart.
  Interventions: Other: TEMPS-A (Temperament Evaluation of Memphis, Pisa, Paris and San Diego Auto-questionnaire)

INTERVENTIONS:
Other: TEMPS-A (Temperament Evaluation of Memphis, Pisa, Paris and San Diego Auto-questionnaire) — Participants filled out the TEMPS-A survey at their first visit.

SUMMARY:
In this study, the investigators aimed to research the relationship between affective temperament with the severity of the symptoms of nausea and vomiting in early pregnancy. The investigators aimed to assess temperament differences between healthy pregnant women and pregnant women suffering from mild, moderate, and severe hyperemesis gravidarum.

ELIGIBILITY:
Inclusion Criteria:

* To be 16 years or older
* To be at the level of education to understand and answer the survey questions
* To have singleton live pregnancy within the first six weeks of pregnancy according to ultrasound measurement or the level of human chorionic gonadotropine in the blood
* Agreed to participate the study by signing a voluntary informed consent form

Exclusion Criteria:

* History of any medical problems (eg. endocrine, gastrointestinal, cardiovascular, pulmonary system diseases, vertigo)
* Presence of a history of psychiatric disorder (eg. depression, anxiety, bipolar disorder, delirium, eating disorders and other psychotic disorders)
* Multiple pregnancy
* Pregnancy complicating situation (eg. imminent abortion, trophoblastic disease, ectopic pregnancy)
* Presence of a history of regular medication use (Including drug use within the last six months for psychiatric illness)
* To be not at the risk for anxiety disorder or depression according to the result of hospital anxiety and depression scale

Ages: 16 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 252 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
TEMPS-A scale measurement | 1 day
  The participants filled out TEMPS-A survey at their first visit.
PUQE scoring index | 2 months
  The investigators performed this test to subjects three times of session separated by a month

SECONDARY OUTCOMES:
Hospital anxiety and depression scale | 1 day
  Used for excluding patients with the risk of anxiety disorder or depression.

CONTACTS AND LOCATIONS:
Overall Officials: ALI BAHADIRLI, M.D., Principal Investigator — Recruiting
Locations (1):
- Mustafakemalpasa Government Hospital, Bursa, Turkey (Türkiye)

REFERENCES:
- [Result] Verberg MF, Gillott DJ, Al-Fardan N, Grudzinskas JG. Hyperemesis gravidarum, a literature review. Hum Reprod Update. 2005 Sep-Oct;11(5):527-39. doi: 10.1093/humupd/dmi021. Epub 2005 Jul 8. PMID 16006438
- [Result] Gadsby R, Barnie-Adshead AM, Jagger C. A prospective study of nausea and vomiting during pregnancy. Br J Gen Pract. 1993 Jun;43(371):245-8. PMID 8373648
- [Result] Einarson TR, Piwko C, Koren G. Quantifying the global rates of nausea and vomiting of pregnancy: a meta analysis. J Popul Ther Clin Pharmacol. 2013;20(2):e171-83. Epub 2013 Jul 13. PMID 23863575
- [Result] Bashiri A, Neumann L, Maymon E, Katz M. Hyperemesis gravidarum: epidemiologic features, complications and outcome. Eur J Obstet Gynecol Reprod Biol. 1995 Dec;63(2):135-8. doi: 10.1016/0301-2115(95)02238-4. PMID 8903768
- [Result] Fell DB, Dodds L, Joseph KS, Allen VM, Butler B. Risk factors for hyperemesis gravidarum requiring hospital admission during pregnancy. Obstet Gynecol. 2006 Feb;107(2 Pt 1):277-84. doi: 10.1097/01.AOG.0000195059.82029.74. PMID 16449112
- [Result] Flaxman SM, Sherman PW. Morning sickness: adaptive cause or nonadaptive consequence of embryo viability? Am Nat. 2008 Jul;172(1):54-62. doi: 10.1086/588081. PMID 18500939
- [Result] Weigel RM, Weigel MM. Nausea and vomiting of early pregnancy and pregnancy outcome. A meta-analytical review. Br J Obstet Gynaecol. 1989 Nov;96(11):1312-8. doi: 10.1111/j.1471-0528.1989.tb03229.x. PMID 2611170
- [Result] Wegrzyniak LJ, Repke JT, Ural SH. Treatment of hyperemesis gravidarum. Rev Obstet Gynecol. 2012;5(2):78-84. PMID 22866186
- [Result] McCarthy FP, Khashan AS, North RA, Moss-Morris R, Baker PN, Dekker G, Poston L, Kenny LC; SCOPE Consortium. A prospective cohort study investigating associations between hyperemesis gravidarum and cognitive, behavioural and emotional well-being in pregnancy. PLoS One. 2011;6(11):e27678. doi: 10.1371/journal.pone.0027678. Epub 2011 Nov 18. PMID 22125621